CLINICAL TRIAL: NCT04926584
Title: Prospective Trial of Immunotherapy Prior to Resection, Definitive Chemo-radiotherapy, or Palliative Therapy in Patients With Locally Advanced or Oligometastatic Non-small Cell Lung Cancer Without a Primary Curative Option
Brief Title: Prospective Trial of Induction Immunotherapy in Locally Advanced or Oligometastatic NSCLC Without a Primary Curative Option
Acronym: KOMPASSneo
Status: Recruiting | Type: Observational
Sponsor: Klinikum Esslingen (Other)
Responsible Party: Principal Investigator, Martin Faehling, Head of Pneumology, Klinikum Esslingen
Other Study IDs: KOMPASSneo
Record Dates: First submitted 2021-06-09; First posted 2021-06-15 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: immunotherapy, chemoradiotherapy, resection, PD-L1
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: induction therapy — induction immuno-chemotherapy or immunotherapy prior to resection or definitive chemoradiotherapy

SUMMARY:
In a certified lung- cancer center, patients with NSCLC and a potentially curative stage (including patients with oligometastatic disease) are prospectively enrolled if curative treatment (either definitive radio-chemotherapy or resection) cannot be performed due to large tumor size or for functional reasons. For these patients, the multidisciplinary tumor board (MDB) recommends immuno-(chemo)therapy and re-evaluation. Response is assessed radiologically including PET-CT if indicated. After review of the MDB, patients receive either definitive curative treatment or palliative treatment.

DETAILED DESCRIPTION:
In a certified lung- cancer center, patients with NSCLC and a potentially curative stage (including patients with oligometastatic disease) are prospectively enrolled if curative treatment (either definitive radio-chemotherapy or resection) cannot be performed due to large tumor size or for functional reasons (e. g. too large radiation field or functionally inoperable for the required resection). For these patients, the multidisciplinary tumor board (MDB) recommends immuno-(chemo)therapy and re-evaluation. Response is assessed radiologically including PET-CT if indicated. After review of the MDB, patients receive either definitive curative treatment or palliative treatment.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed NSCLC
* histologically or cytologically proven
* stage III - IVA (oligometastatic) by complete staging
* ECOG 0-2
* life expectancy 3 months
* ability to provide written informed consent

Exclusion Criteria:

* primary resectability
* primary definitive chemoradiotherapy feasible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with locally advanced or oligometastatic NSCLC (stage IIIA - IVA) wae elegible if curative treatment (either resection or chemoradiotherapy is not possible for anatomical or functional reasons
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-12-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
patients completing definitive therapy | 1 year
  proportion of patients completing definitive therapy

SECONDARY OUTCOMES:
complete or partial radiologic response | 1 year
  proportion of patients who achieved complete or partial radiologic response
local downstaging | 1 year
  proportion who achieved local downstaging
complete metabolic response | 1 year
  proportion who achieved complete metabolic response
overall survival (OS) | 5 years
  overall survival (OS)
event-free survival (EFS) | 5 years
  event-free survival (EFS)

CONTACTS AND LOCATIONS:
Locations (1):
- Klinikum Esslingen, Esslingen am Neckar, Germany

IPD SHARING:
Plan to Share IPD: No